CLINICAL TRIAL: NCT03673410
Title: A Randomized Study of Robotic Versus Laparoscopic Techniques for Revisional Bariatric Surgery
Brief Title: Robotic Versus Laparoscopic Techniques for Revisional Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Robotic revisional surgery
Record Dates: First submitted 2018-09-05; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Bariatric Surgery; Robotic Surgery

STUDY DESIGN:
Intervention Model Description: We will randomise 60 patients between robotic (30 patients) and laparoscopic revisional bariatric surgery (30 patients) to evaluate those procedures in terms of perioperative safety, weight loss and comorbidity resolution.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Once consent has been signed, the patient will be assigned to any of the two groups, using a computer-based randomization on REDCap and the patient will be assigned to the corresponding study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic revisional bariatric surgery (Active Comparator): Patients requiring revisional bariatric surgery will be treated with a standard of care laparoscopic procedure.
  Interventions: Procedure: Laparoscopic bariatric surgery - revisional
- Robotic revisional bariatric surgery (Experimental): Patients requiring revisional bariatric surgery will be treated with the same procedure but performed robotically.
  Interventions: Procedure: Robotic bariatric surgery - revisional

INTERVENTIONS:
Procedure: Robotic bariatric surgery - revisional — Using robotic techniques during any revesional bariatric surgery
  Arms: Robotic revisional bariatric surgery
Procedure: Laparoscopic bariatric surgery - revisional — Using laparoscopic techniques during any revesional bariatric surgery
  Arms: Laparoscopic revisional bariatric surgery

SUMMARY:
Obesity has become a significant health problem in Canada. When conservative efforts to lose weight fail, bariatric surgical procedures are often considered. Today, the most common bariatric procedures in North America are Laparoscopic Roux-en-Y gastric bypass (LRYGB) and Laparoscopic Sleeve Gastrectomy (LSG).

For many reasons, an initial bariatric procedure may require surgical revision. Some reasons include weight regain, failed weight loss or other acute and chronic complications not related to weight loss. In these cases, it may be indicated that a procedure be reversed inor converted to another type of bariatric procedure. Regardless of the planned intervention, revisional surgery is always more difficult than the initial procedure mainly due to surgical scarring and altered anatomy. Though revisional bariatric surgery has been shown to be safe, our hope is to improve the safety profile by utilizing robotic surgery. Robotic surgery can facilitate more complex procedures by providing superior imaging and freedom of movement during the procedure.

The aim of our study is to evaluate prospectively the outcomes of robotic compared to laparoscopic revisional bariatric surgery in terms of perioperative outcomes such as complication rates, operative time and readmissions as well as weight loss/comorbidity resolution (diabetes, hypertension, sleep apnea) where applicable.

DETAILED DESCRIPTION:
Revisional bariatric surgery is becoming increasingly commonplace in surgical practices. Approximately 10-25% of patients bariatric surgery will require a revisional procedure at some point after their initial operation. A conversion from one procedure to another can take place as part of a planned two-step procedure or due to failed weight loss or weight regain after the initial procedure. Furthermore, patients can require revision due to other acute and chronic complications such as marginal ulcers, stenosis and nausea/vomiting. Though these procedures are generally successful in their intended goal, it is been reported that complication rates are higher after revision surgery the primary bariatric procedures. Despite this, few studies have explored methods of increasing safety for revisional bariatric surgery.

Robotic surgery is a tool that could potentially aid in the safety of revisional bariatric surgery. Specific to bariatric surgery, the major strengths of robotic surgery is in facilitating more complex surgical steps, such as a hand-sewn gastrojejunostomy, and providing superior imaging and freedom of movement compared to traditional laparoscopy. While these advantages may not confer major benefits in primary bariatric surgery, revisional bariatric surgery often requires hand-sewn anastomoses in anatomical locations made more difficult by previous surgical scarring and altered anatomy. This may also translate into a long-term clinical and economic benefit which could offset the costs of robotics.

Despite this potential, there have been relatively few studies that have investigated the use of robotic assistance during revisional bariatric surgery and almost none with long-term data. Furthermore, there is a paucity of high-quality research demonstrating any intervention that increases safety during revisional bariatric surgery, including robotics. Considering the current and future demand revisional bariatric surgery, there is a large potential role for any interventions that can increase safety during these operations.

Aim:

The aim of our study is to prospectively evaluate the difference between robotic and laparoscopic revisional bariatric surgery in major surgical outcomes and metabolic outcomes, where applicable.

Study Population:

Patients seen in the bariatric clinic and judged to be potential candidates for revisional of bariatric surgery will be screened as potential candidates for this study.

Inclusion Criteria

Participants must meet all of the following inclusion criteria:

* The subject previously met National Institutes of Health criteria for bariatric surgery11 and received a bariatric surgical procedure.
* The subject is under consideration to undergo a revisional bariatric procedure after for failed sustained weight loss, weight regain or other chronic issues requiring revision.
* The subject is able and willing to give written consent
* The subject must be 18-70 years of age
* The subject must be willing and able to participate in the study procedures and to understand and sign the informed consent

Exclusion criteria

Participants who meet any of the following criteria at the time of the baseline visit are NOT eligible to be enrolled in this study:

* The subject has a contraindication to general anesthesia
* The revision does not occur within the first 90 days of the initial bariatric procedure
* The subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* The subject is a pregnant or lactating female (Women of child bearing potential must take a pregnancy test prior to surgery)
* The subject has an history of alcohol abuse (>30 g/day in men or >20 g/day in women)
* Any subject who is considered to be part of a vulnerable population (e.g. prisoners or those with psychological concerns or those without sufficient mental capacity)
* The subject is unable or unwilling to comply with the study requirements or follow-up schedule
* The subject has conditions which, in the opinion of the investigator, will not be appropriate for the study (e.g. severe cardiovascular disease, history of gastrointestinal (GI) malignancy, history of upper GI surgery, open cholecystectomy, history of intestinal surgery, immunosuppression, or non-ambulatory)
* The subject has an estimated life expectancy of less than 6 months

Methodology

All patients will have routine pre-operative bariatric clinic assessment. This includes, among other things, complete medical history and physical exam, endoscopy, abdominal ultrasound and blood tests. This involves the nurse, surgeon and internal medicine doctor that will evaluate the patient regarding co-morbidities.

A prospective study will be able to start in January 2019 and will have a single surgeon performing robotic revisional bariatric surgery at St. Joseph Healthcare. Robotic revisional bariatric surgery will be performed according to the National Institutes of Health, as well as the American College of Surgeons (ACS) and the American Society for Metabolic and Bariatric Surgery (ASMBS) guidelines. This study will include patients over 18 years-old who have previously undergone bariatric surgery and a require revisional procedure. The investigators will collect demographic data related to the patient such the age, gender, weight, height, BMI, comorbidities such as hypertension, sleep apnea, hypertriglyceridemia, hypercholesterolemia, type 2 diabetic (with or without insulin therapy). The investigators will assess the operative time, the immediate postoperative complication rate according to Dindo-Clavien classification, the mean length of hospital stay, the thirty-day readmission rate, the thirty-day reoperation rate and the long-term reintervention rate. Follow-up of the patients at 6 months, 1, 3 and 5 years, will be conducted as per usual through the bariatric clinic where secondary outcomes will be assessed.

The investigators will randomise 60 patients between robotic (30 patients) and laparoscopic revisional bariatric surgery (30 patients) to evaluate those procedures in terms of perioperative safety, weight loss and comorbidity resolution.

Consent:

Patients will be approached for consent during their preoperative evaluation visits at the Bariatric Clinic. Members of the study team will explain the study to the patient, answer questions and will explain the informed consent form. Once all questions have been answered to the patient's satisfaction, the patient will be asked to provide written informed consent.

Randomization:

Once consent has been signed, the patient will be assigned to any of the two groups, using a computer-based randomization on REDCap and the patient will be assigned to the corresponding study arm.

Screening:

The patients will have all screening done before consent is signed.

Potential risk:

Potential risks of this study are related to surgery. The patient should not have any increased risk when assigned to the study group robotic vs standard surgical treatment.

Safety:

Safety will be assessed on an ongoing basis by the Principal Investigator. All adverse events will be evaluated as they occur by the Principal Investigator to determine the study continuance and to make any modifications to the procedure when necessary.

Assessment of outcomes

Primary Outcomes

Surgical Complications:

These will be defined by the Clavien-Dindo classification and our primary outcome will be long-term complications higher than grade III:

Grade III: Requiring surgical, endoscopic or radiological intervention Grade III-a: intervention not under general anesthesia Grade III-b: intervention under general anesthesia Grade IV: Life-threatening complication (including CNS complications)‡ requiring IC/ICU-management Grade IV-a: single organ dysfunction (including dialysis) Grade IV-b: multi organ dysfunction Grade V: Death of a patient

Long-term reintervention rate:

Reinterventions for chronic surgical complications will be assessed through the bariatric clinic. Only complications related to the procedure, such as therapeutic endoscopy or reoperation will be counted.

Secondary Outcomes

Hypertension:

The presence and remission of hypertension will be diagnosed by the definitions suggested in 2003 by the seventh report of the Joint National Committee (JNC 7) and are based upon the average of two or more properly measured readings at each of two or more office visits after an initial screen:

* Normal blood pressure: systolic <120 mmHg and diastolic <80 mmHg
* Prehypertension: systolic 120 to 139 mmHg or diastolic 80 to 89 mmHg (see "Prehypertension")
* Hypertension:

  * Stage 1: systolic 140 to 159 mmHg or diastolic 90 to 99 mmHg
  * Stage 2: systolic ≥160 mmHg or diastolic ≥100 mmHg

Type 2 diabetes:

The presence and remission of type 2 diabetes will be diagnosed according to the American Diabetes Association's current criteria:

1. A1C ≥6.5 percent, OR
2. FPG ≥126 mg/dL (7.0 mmol/L), OR
3. Two-hour plasma glucose ≥200 mg/dL (11.1 mmol/L) during an OGTT, OR
4. In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥200 mg/dL (11.1 mmol/L).

Post-surgical evaluation:

All patients will undergo the standard bariatric postoperative evaluation including:

• Appointments with the bariatric team (surgeon, internist, nurse, dietitian, social worker and psychologist) at 1 week, 1 month, 3 months, 6 months, 9 months, 1 year, and then on a yearly basis until at least 5 years after date of surgery.

Statistical analysis:

Descriptive statistics (means, medians, standard deviations) will be used to characterize the patient population where applicable. Chi square was used to analyze dichotomous patient variables such as adverse events while continuous variables were analysed using T-tests.

Our primary outcome will be any reintervention, readmission or grade 2, 3, 4 or 5 complication over the entire period of the study. Interim analysis will be done at years 1 and 3. Participants will be followed followed for the 5 years postoperatively. This study is designed to assess a 50% reduction in time to the primary outcome, with p <0.05 and 80% power (assuming a major complication/reintervention rate of approximately 20% in the literature).

The primary outcome will be evaluated using a hazard ratio and time-to-event analysis. Kaplan-Meier curves will created for both groups and compared in a univariable manner using the log rank test. Two Cox models will then created to assess the hazard ratio between the treatment and control groups. The first will be a univariable model using treatment as the only variable. A second, multivariable will be created to ascertain the effect of the treatment after adjustment for important variable.

Our secondary metabolic outcomes will be assessed using a log transformed generalized linear model with robust confidence intervals for binary and continuous outcomes, where appropriate. For binary outcomes, this provides the risk ratios for the effect estimate of robotic vs laparoscopic approaches. Two regression models will be created to assess the differneces between the treatment and control groups. The first will be a univariable model using treatment as the only variable. A second, multivariable was created to ascertain the effect of the treatment after adjustment for important variables that may not have been balanced during randomization.

Monte Carlo Markov Chain estimation will be used for the regression models with 100,000 iterations after a 5,000 iteration burn-in. All chains were examined for convergence. Statistical significance was set at p < 0.05. Data were analyzed using Stata (StataCorp version 12.1; College Station, TX) and MLwiN (Version 2.26; Centre for Multilevel Modelling, University of Bristol).

ELIGIBILITY:
Inclusion Criteria:

* The subject previously met National Institutes of Health criteria for bariatric surgery11 and received a bariatric surgical procedure.
* The subject is under consideration to undergo a revisional bariatric procedure after for failed sustained weight loss, weight regain or other chronic issues requiring revision.
* The subject is able and willing to give written consent
* The subject must be 18-70 years of age
* The subject must be willing and able to participate in the study procedures and to understand and sign the informed consent

Exclusion Criteria:

* The subject has a contraindication to general anesthesia
* The revision does not occur within the first 90 days of the initial bariatric procedure
* The subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* The subject is a pregnant or lactating female (Women of child bearing potential must take a pregnancy test prior to surgery)
* The subject has an history of alcohol abuse (>30 g/day in men or >20 g/day in women)
* Any subject who is considered to be part of a vulnerable population (e.g. prisoners or those with psychological concerns or those without sufficient mental capacity)
* The subject is unable or unwilling to comply with the study requirements or follow-up schedule
* The subject has conditions which, in the opinion of the investigator, will not be appropriate for the study (e.g. severe cardiovascular disease, history of gastrointestinal (GI) malignancy, history of upper GI surgery, open cholecystectomy, history of intestinal surgery, immunosuppression, or non-ambulatory)
* The subject has an estimated life expectancy of less than 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Short term complication rate | 30 days from surgery
  Any complication - Complication will be defined by the Clavien-Dindo classification and our primary outcome will be long-term complications higher than grade III. These will include leaks and bleeds.
  Only complications related to the procedure, such as therapeutic endoscopy or reoperation will be counted.
  3)
Readmission | 30 days from surgery
  Readmission to the center within 30 days of the original procedure
Long-term reintervention | 5 years
  Reinterventions for chronic surgical complications (such as stricture) will be assessed through the bariatric clinic.
  Only reintenrtventinos related to the original procedure will be counted.

SECONDARY OUTCOMES:
Weight loss in kgs | 1, 3, 5 years
  This is the change in weight from the date of operation 2) 3) 4) 5) Sleep apnea (binary, defined as no need for CPAP)
BMI change (in kg/m2) | 1, 3 and 5 years
  This is the change in BMI from the date of operation
Diabetes resolution | 1, 3 and 5 years
  This is a binary outcome relating to the resolution of diabetes from baseline defined as no need for medication
Hypertension resolution | 1, 3, and 5 years
  This is a binary outcome relating to the resolution of hypertension from baseline defined as no need for medication
Sleep apnea resolution | 1, 3, and 5 years
  This is a binary outcome relating to the resolution of sleep apnea from baseline defined as no need for medication

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hong, MD Msc, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No